CLINICAL TRIAL: NCT04154072
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of 36 Weeks of Treatment With NLY01 in Early-stage Parkinson's Disease
Brief Title: A Clinical Study of NLY01 in Patient's With Early Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuraly, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLY01-PD-1
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NLY01 (2.5 mg) (Active Comparator): NLY01 2.5 mg injection
  Interventions: Drug: NLY01
- NLY01 (5.0 mg) (Active Comparator): NLY01 5.0 mg injection
  Interventions: Drug: NLY01
- Vehicle (Placebo Comparator): inactive drug, injection
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: NLY01 — exenatide and polyethylene glycol (PEG)
  Arms: NLY01 (2.5 mg); NLY01 (5.0 mg)
Drug: Vehicle — Saline (Sodium Chloride)
  Arms: Vehicle

SUMMARY:
This is a phase 2 study designed to assess the safety, tolerability and efficacy of NLY01 in subjects with early untreated Parkinson's disease (PD). Evidence suggests NLY01, a pegylated form of exenatide, may be beneficial in PD and is being developed as a potential treatment for neurodegenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with Parkinson's disease according to UK Parkinson's Disease Society Brain Bank Clinical Diagnostic criteria or Movement Disorder Society Research Criteria
* Patients with Parkinson's disease according to protocol specified scale assessments
* DaTscan consistent with diagnosis of Parkinson's Disease
* Men or women 30 to 80 years of age

Exclusion Criteria:

* Diagnosis of secondary or atypical parkinsonism
* Prior use of dopaminergic treatment or MAO-B inhibitors for more than 28 days
* Medical or recreational use of marijuana or THC-containing compounds within 3 months of screening visit
* Pregnant or planning to become pregnant
* Metabolic, surgical, psychiatric or laboratory abnormality that would interfere with study compliance or safety in the judgment of the investigator

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale in combined score of Parts II and III from baseline to 36 weeks | 36 weeks
  This is the Unified Parkinson's Disease Rating Scale assessment (MDS-UPDRS). The investigator will assess II and III components of the Unified Parkinson's Disease Rating Scale. The Unified Parkinson's Disease Rating Scale Part II assesses motor aspects of experiences of daily living. The Unified Parkinson's Disease Rating Scale Part III assesses motor signs of Parkinson's Disease.
  The Unified Parkinson's Disease Rating Scale is a widely used assessment to quantify the signs and symptoms of Parkinson's Disease. Each subscale has 0-4 ratings, where 0=normal, 1=slight, 2=mild, 3=moderate and 4=severe. The scale is completed by the investigator and scores are derived from clinician and subject input to allow the assessment of symptomatic worsening and improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Lee, Study Director — Neuraly, Inc.
Locations (61):
- United States (60):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center - Barrow Neurological Institute, Phoenix, Arizona
  - Movement Disorders Center, Scottsdale, Arizona
  - Mayo Clinic Arizona, Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, Irvine, Irvine, California
  - Keck School of Medicine of USC/University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Center for Neurotherapeutics, Los Angeles, California
  - SC3 Research, Pasadena, California
  - University of California Davis Health, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Rocky Mountain Movement Disorder Center, Englewood, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorder Center, Boca Raton, Florida
  - Nova Clinical Research, Bradenton, Florida
  - University of Florida, Gainesville, Florida
  - Infinity Clinical Research, Hollywood, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Visionary Investigators Network, Miami, Florida
  - University of Miami, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - University of South Florida, Tampa, Florida
  - Charter Research, Winter Park, Florida
  - Augusta University, Augusta, Georgia
  - NeuroStudies, Decatur, Georgia
  - Northwestern Medical Group Neurology Clinic, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - SIU Medicine, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland, Neurology Ambulatory Center, Maryland Parkinson's Disease and Movement Disorder Center, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital Clinical Trials Pharmacy, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - University of Minnesota Delaware Clinical Research Unit, Minneapolis, Minnesota
  - Neurology Specialists of Monmouth County, West Long Branch, New Jersey
  - NYU Langone Medical Center, The Marlene and Paolo Fresco Institute for Parkinson's and Movement Disorders, New York, New York
  - Neurological Institute, Columbia University Medical Center, New York, New York
  - UNC CTRC, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Raleigh Neurology, Raleigh, North Carolina
  - Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Toledo, Gardner-McMaster Parkinson Center, Toledo, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McGarry A, Rosanbalm S, Leinonen M, Olanow CW, To D, Bell A, Lee D, Chang J, Dubow J, Dhall R, Burdick D, Parashos S, Feuerstein J, Quinn J, Pahwa R, Afshari M, Ramirez-Zamora A, Chou K, Tarakad A, Luca C, Klos K, Bordelon Y, St Hiliare MH, Shprecher D, Lee S, Dawson TM, Roschke V, Kieburtz K. Safety, tolerability, and efficacy of NLY01 in early untreated Parkinson's disease: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2024 Jan;23(1):37-45. doi: 10.1016/S1474-4422(23)00378-2. PMID 38101901